CLINICAL TRIAL: NCT04122898
Title: Effect of Pelvic Floor Muscles Training on Symptoms, Bother and Amount of Stress Urinary Incontinence in Female Gymnasts, Team Gymnasts and Cheerleaders. An Assessor Blinded Randomized Controlled Trial
Brief Title: Pelvic Floor Muscle Training in Gymnasts With Stress Urinary Incontinence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to covid-19
Sponsor: Norwegian School of Sport Sciences (Other)
Responsible Party: Principal Investigator, Kari Bø, Professor, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KLS2019
Record Dates: First submitted 2019-10-04; First posted 2019-10-10 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Urinary Incontinence; Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Three months home-based PFM training program with weekly follow-up by a physiotherapist
  Interventions: Other: Pelvic Floor Muscle Training
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Other: Pelvic Floor Muscle Training — The intervention will consist of a home-based PFM training program with weekly follow-up by phone by a physiotherapist. Before commencing PFM training, the gymnasts in the intervention group will have an individual session with a physiotherapist including thorough teaching on how to perform a correct PFM contraction (inward lift of the pelvic floor assessed with suprapubic 2D ultrasound) and instructions on how to perform the training program. The athletes will be offered at least one individual follow-up session with the same physiotherapist during the intervention period. The program will consist of 3 sets of 8-12 maximum contractions per day. An electronic app (Athlete monitoring) will be used to assess adherence to the program. The athletes will be asked to register their training sessions in a personal account. A reminder to adhere to the program will be sent by phone. The training period will be 3 months and the exercises will take approximately 10 minutes per day to perform.
  Other Names: Pelvic Floor Muscle Training in Elite Gymnasts
  Arms: Intervention Group

SUMMARY:
There is a high prevalence of urinary incontinence (UI) among female athletes participating in high impact sports, such as artistic gymnastics, trampoline jumping and ball games. UI is defined as "the complaint of involuntary loss of urine". Stress urinary incontinence (SUI) is the most common type of UI and is defined as "the complaint of involuntary loss of urine on effort or physical exertion (e.g. sporting activities), or or sneezing or coughing". Urinary leakage during sport activities may affect the athletes' performance, cause bother, frustration and embarrassment and furthermore lead to avoidance and cessation of sport activities. Pelvic floor muscle (PFM) training is highly effective in treating SUI in the general female population. However, evidence of the effect of PFM training in elite athletes in high impact sports is sparse.

The purpose of this assessor-blinded randomized controlled trial (RCT) is to assess the effect of PFM training on symptoms, bother and amount of SUI in female artistic gymnasts, team gymnasts and cheerleaders.

DETAILED DESCRIPTION:
BACKGROUND:

Physical activity and exercise have well-known beneficial effects on several physical and psychological health outcomes. However, it has been proposed that regular participation in physical activity and exercise may lead to greater risk of developing pelvic floor dysfunctions (PFD) in women. The pelvic floor consists of muscles, fascia and ligaments and forms a hammock-like support at the base of the abdomino-pelvic cavity. The function of the pelvic floor is to provide support to the pelvic organs (the bladder, urethra, vagina, uterus and rectum) and to counteract all increases in intra-abdominal pressure and ground reactions forces during daily activities. Additionally, the pelvic floor facilitates intercourse, vaginal birth, storage of stool and urine and voluntary defecation and urination. A dysfunctional pelvic floor can lead to urinary and anal incontinence, pelvic organ prolapse, sexual problems and chronic pain syndromes. UI is the most common PFD, defined as "the complaint of involuntary loss of urine". SUI, urgency urinary incontinence (UUI) and mixed urinary incontinence (MUI) are common subtypes of UI. In women, SUI accounts for approximately half of all incontinence types and is defined as "the complaint of involuntary loss of urine on effort or physical exertion (e.g. sporting activities), or on sneezing or coughing". UUI is defined as the "complaint of involuntary loss of urine associated with urgency" and MUI as "complaints of both stress and urgency urinary incontinence".

High prevalence rates of UI among both parous and nulliparous female athletes and exercisers have been reported in several cross-sectional studies. The prevalence rates varies between 0-80% with the highest prevalence found in high impact sports such as trampoline jumping, gymnastics and ball games. Leakage during sport activities may affect the athletes' performance and cause bother, frustration and embarrassment. Some athletes have reported that UI issues have also led to avoidance or cessation of sport or exercise.

To date, there is level 1 evidence and grade A recommendation for PFM training alone to be first line treatment for SUI, MUI and pelvic organ prolapse in the general female population. In addition, PFM training is highly effective as primary prevention; pregnant continent women who exercise the PFM are at 62% less risk of UI in late pregnancy and 29% less risk of UI 3-6 months postpartum. Evidence of the effect of PFM training in athletes or strenuous exercisers is sparse.

In one study on female soldiers and two small case series in female athletes and exercisers, PFM training led to reduced symptoms of UI. However, none of these studies included a non-treated control group and the internal validity is therefore low. To our knowledge, only one RCT has assessed effects of PFM training on SUI in athletes. Female volleyball players (n=16) who followed a PFM training program had significant improvements of SUI compared to a control group (n=16).

Based on today's knowledge we do not know whether PFM training is effective in elite athletes exposed to excessive impact in sports including elements of acrobatics and jumping. Given the high impact on the pelvic floor in these athletes, it is presumed that they need much better pelvic floor muscle function than non-exercisers. On the other hand, elite athletes are highly motivated for regular training. Strength training of the PFM, if proven effective, may be easily incorporated in their basic training regimens both as prevention and treatment strategies of SUI.

AIMS:

The aim of this RCT is to assess the effect of PFM training on symptoms, bother and amount of SUI among female artistic gymnasts, team gymnasts and cheerleaders.

STUDY DESIGN AND METHODS:

A cross-sectional study will be conducted to assess prevalence of SUI among female artistic gymnasts, team gymnasts and cheerleaders from 12 years of age competing on high national levels in Norway. Athletes reporting symptoms of SUI will be asked to participate in the RCT.

The study is an assessor-blinded RCT evaluating the effect of PFM training on SUI in elite female gymnasts, team gymnasts and cheerleaders. At baseline, all athletes will perform a pad weight-test, measuring the amount of leakage during gymnastic and acrobatic activities. In addition, the athletes will respond to a standardized questionnaire, measuring self-reported symptoms of UI and bother. The athletes will be randomly assigned to either a PFM training group (EG) or a control group (CG) with no intervention. The intervention consists of a daily home-based PFM training program with weekly follow-up by a physiotherapist. After a three-months intervention period, all athletes will perform a post-test including the same previous mentioned outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* female artistic gymnasts, team gymnasts and cheerleaders
* eligible to compete in the Norwegian National Championship or competitions of higher levels
* > 12 years of age
* total score on ICIQ-UI-SF of >3
* positive pad weight-test: >1 gram of leakage
* self-reported SUI with ICIQ-UI-SF (urinary leakage during physical activity, exercise, sneezing or coughing)

Exclusion Criteria:

* history of pregnancy, pelvic surgery, pelvic trauma, inflammatory bowel diseases or respiratory diseases/symptoms
* male gymnasts
* < 12 years of age
* not eligible to competed in the Norwegian National Championship or competitions of higher levels
* athletes who are unable to correctly contract the PFM, examined by suprapubic transabdominal 2D ultrasound

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2020-08-19 (Actual)

PRIMARY OUTCOMES:
Pad-weight Stress Test for Stress Urinary Incontinence | Change from baseline pad-test at three months
  The test will be modified from the descriptions by Mørkved & Bø, Eliasson, Larsson & Mattson and Ferreira et al. The athletes will be requested to void 30 minutes before the test, to drink 0.5 liter of water and thereafter not empty their bladder. A pre-weighted pad will be applied, and the athletes will perform a 10 minutes intensive warm-up followed by 5 minutes of high impact gymnast- or cheerleading routines.

SECONDARY OUTCOMES:
The International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI-SF) | Change in total score from baseline at three months
  A reliable and valid questionnaire assessing self-reported prevalence, amount of leakage, bother and type of UI. A change in ICIQ-UI-SF score of 1.58 points will be considered as between-treatment minimum important difference.
Patient Global Impression of Improvement (PGI-I) Scale | Post-test after a 3-months intervention period
  The gymnasts will be asked to rate their perceived change of the condition. A validated 7-point scale with response choices ranging from "very much better" to "very much worse" will be used.
Self-Efficacy Scale for Practicing Pelvic Floor Exercises (SESPPFE) | At baseline in both groups. Athletes in the intervention group will also be asked to answer the questionnaire again within the first month of the intervention period.
  The gymnasts will be asked to rate their self-efficacy (from 0-100) on 16 different items regarding PFM training. The scale have been tested to have good internal consistency (α = 0.92) and acceptable reliability (rho = 0.89).

CONTACTS AND LOCATIONS:
Overall Officials: Kari Bø, PhD, Study Chair — Norwegian School of School of Sport Sciences
Locations (1):
- Norwegian School of Sport Sciences, Department of Sport Medicine, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piercy KL, Troiano RP. Physical Activity Guidelines for Americans From the US Department of Health and Human Services. Circ Cardiovasc Qual Outcomes. 2018 Nov;11(11):e005263. doi: 10.1161/CIRCOUTCOMES.118.005263. No abstract available. PMID 30571339
- [Background] Ruiz-Zapata, A. M., Feola, A. J., Heesakkers, J., de Graaf, P., Blaganje, M., & Sievert, K. D. (2018). Biomechanical Properties of the Pelvic Floor and its Relation to Pelvic Floor Disorders. European Urology Supplements, 17(3), 80-90.
- [Background] Bump RC, Norton PA. Epidemiology and natural history of pelvic floor dysfunction. Obstet Gynecol Clin North Am. 1998 Dec;25(4):723-46. doi: 10.1016/s0889-8545(05)70039-5. PMID 9921553
- [Background] Milsom, I., Altman, D., Cartwright, R., Lapitan, M. C. M., Nelson, R., Sjöström, S., & Tikkinen, K. A. O. (2017). Epidemiology of urinary incontinence (UI) and other lower urinary tract symptoms (LUTS), pelvic organ prolapse (POP) and anal (AI) incontinence. In P. C. Abrams, L.; Wagg, A.; Wein, A. (Ed.), Incontinence (Vol. 1, pp. 1-141). Tokyo: 6th International Consultation on Incontinence.
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Int Urogynecol J. 2010 Jan;21(1):5-26. doi: 10.1007/s00192-009-0976-9. Epub 2009 Nov 25. PMID 19937315
- [Background] Bø, K. (2015). Pelvic floor dysfunction, prevention and treatment in elite athletes. In K. Bø, B. Berghmans, S. Mørkved, & M. Van Kampen (Eds.), Evidence based Physical Therapy for the Pelvic Floor - Bridging science and clinical practice (pp. 397-407). Edinburgh London New York Oxford Philadelphia St Louis Sydney Toronto: Elsevier Churchilll Livingstone.
- [Background] de Mattos Lourenco TR, Matsuoka PK, Baracat EC, Haddad JM. Urinary incontinence in female athletes: a systematic review. Int Urogynecol J. 2018 Dec;29(12):1757-1763. doi: 10.1007/s00192-018-3629-z. Epub 2018 Mar 19. PMID 29552736
- [Background] Nygaard IE, Shaw JM. Physical activity and the pelvic floor. Am J Obstet Gynecol. 2016 Feb;214(2):164-171. doi: 10.1016/j.ajog.2015.08.067. Epub 2015 Sep 6. PMID 26348380
- [Background] Jacome C, Oliveira D, Marques A, Sa-Couto P. Prevalence and impact of urinary incontinence among female athletes. Int J Gynaecol Obstet. 2011 Jul;114(1):60-3. doi: 10.1016/j.ijgo.2011.02.004. Epub 2011 May 14. PMID 21571270
- [Background] Nygaard IE, Thompson FL, Svengalis SL, Albright JP. Urinary incontinence in elite nulliparous athletes. Obstet Gynecol. 1994 Aug;84(2):183-7. PMID 8041527
- [Background] Poswiata A, Socha T, Opara J. Prevalence of stress urinary incontinence in elite female endurance athletes. J Hum Kinet. 2014 Dec 30;44:91-6. doi: 10.2478/hukin-2014-0114. eCollection 2014 Dec 9. PMID 25713669
- [Background] Carls C. The prevalence of stress urinary incontinence in high school and college-age female athletes in the midwest: implications for education and prevention. Urol Nurs. 2007 Feb;27(1):21-4, 39. PMID 17390923
- [Background] Eliasson K, Edner A, Mattsson E. Urinary incontinence in very young and mostly nulliparous women with a history of regular organised high-impact trampoline training: occurrence and risk factors. Int Urogynecol J Pelvic Floor Dysfunct. 2008 May;19(5):687-96. doi: 10.1007/s00192-007-0508-4. Epub 2008 Jan 26. PMID 18224267
- [Background] Hagovska M, Jan S, Bukova A, Horbacz A, Drackova D, Svihrova V, Kraus L. Correction: Prevalence of Urinary Incontinence in Females Performing High-Impact Exercises. Int J Sports Med. 2017 Mar;38(3):e1. doi: 10.1055/s-0043-120578. Epub 2018 Jan 22. No abstract available. PMID 29359297
- [Background] Dumoulin C, Cacciari LP, Hay-Smith EJC. Pelvic floor muscle training versus no treatment, or inactive control treatments, for urinary incontinence in women. Cochrane Database Syst Rev. 2018 Oct 4;10(10):CD005654. doi: 10.1002/14651858.CD005654.pub4. PMID 30288727
- [Background] Woodley SJ, Boyle R, Cody JD, Morkved S, Hay-Smith EJC. Pelvic floor muscle training for prevention and treatment of urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2017 Dec 22;12(12):CD007471. doi: 10.1002/14651858.CD007471.pub3. PMID 29271473
- [Background] Da Roza T, Brandao S, Mascarenhas T, Jorge RN, Duarte JA. Volume of training and the ranking level are associated with the leakage of urine in young female trampolinists. Clin J Sport Med. 2015 May;25(3):270-5. doi: 10.1097/JSM.0000000000000129. PMID 25010151
- [Background] Rivalta M, Sighinolfi MC, Micali S, De Stefani S, Torcasio F, Bianchi G. Urinary incontinence and sport: first and preliminary experience with a combined pelvic floor rehabilitation program in three female athletes. Health Care Women Int. 2010 May;31(5):435-43. doi: 10.1080/07399330903324254. PMID 20390664
- [Background] Sherman RA, Davis GD, Wong MF. Behavioral treatment of exercise-induced urinary incontinence among female soldiers. Mil Med. 1997 Oct;162(10):690-4. PMID 9339085
- [Background] Ferreira, S., Ferreira, M., Carvalhais, A., Santos, P. C., Rocha, P., & Brochado, G. (2014). Reeducation of pelvic floor muscles in volleyball athletes. Rev Assoc Med Bras, 60(5), 428-433.
- [Background] Morkved S, Bo K. The effect of postpartum pelvic floor muscle exercise in the prevention and treatment of urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 1997;8(4):217-22. doi: 10.1007/BF02765817. PMID 9449300
- [Background] Eliasson K, Larsson T, Mattsson E. Prevalence of stress incontinence in nulliparous elite trampolinists. Scand J Med Sci Sports. 2002 Apr;12(2):106-10. doi: 10.1034/j.1600-0838.2002.120207.x. PMID 12121428
- [Background] Avery K, Donovan J, Peters TJ, Shaw C, Gotoh M, Abrams P. ICIQ: a brief and robust measure for evaluating the symptoms and impact of urinary incontinence. Neurourol Urodyn. 2004;23(4):322-30. doi: 10.1002/nau.20041. PMID 15227649
- [Background] Nystrom E, Sjostrom M, Stenlund H, Samuelsson E. ICIQ symptom and quality of life instruments measure clinically relevant improvements in women with stress urinary incontinence. Neurourol Urodyn. 2015 Nov;34(8):747-51. doi: 10.1002/nau.22657. Epub 2014 Aug 22. PMID 25154378
- [Background] Yalcin I, Bump RC. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol. 2003 Jul;189(1):98-101. doi: 10.1067/mob.2003.379. PMID 12861145
- [Background] Sacomori C, Cardoso FL, Porto IP, Negri NB. The development and psychometric evaluation of a self-efficacy scale for practicing pelvic floor exercises. Braz J Phys Ther. 2013 Jul-Aug;17(4):336-42. doi: 10.1590/S1413-35552013005000104. Epub 2013 Aug 30. English, Portuguese. PMID 24072223